CLINICAL TRIAL: NCT02131662
Title: A Randomized, Parallel-group, Double-blind, Placebo Controlled, Multi-center Study to Assess the Efficacy and Safety of Different Doses of BAY1002670 in Subjects With Uterine Fibroids Over 3 Months
Brief Title: Bay1002670, Fibroids, Safety and Efficacy EU,US,Can, Jap
Acronym: ASTEROID 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15788; 2013-003945-40 (EudraCT Number)
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Leiomyoma
Keywords: Uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VPR 4 mg (Experimental)
  Interventions: Drug: BAY1002670
- VPR 2 mg (Experimental)
  Interventions: Drug: BAY1002670
- VPR 1 mg (Experimental)
  Interventions: Drug: BAY1002670
- VPR 0.5 mg (Experimental)
  Interventions: Drug: BAY1002670
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1002670 — Subjects received 4 milligram (mg) Vilaprisan (VPR) tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
  Arms: VPR 4 mg
Drug: BAY1002670 — Subjects received 2 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
  Arms: VPR 2 mg
Drug: BAY1002670 — Subjects received 1 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
  Arms: VPR 1 mg
Drug: BAY1002670 — Subjects received 0.5 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
  Arms: VPR 0.5 mg
Drug: Placebo — Subjects received matching placebo tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
  Arms: Placebo

SUMMARY:
The study is performed to assess the efficacy and safety of different doses of BAY1002670 in subjects with uterine fibroids. The dose-response relationship will be evaluated. Further, the study aims to establish a population pharmacokinetic/pharmacodynamic relationship for BAY1002670 in subjects with uterine fibroids. To assess the efficacy of BAY1002670 the interchangeability of menstrual pictogram and alkaline hematin method for the judgement of menstrual blood loss will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Diagnosis of uterine fibroid(s) documented by transvaginal or abdominal ultrasound at screening with at least 1 fibroid with largest diameter 3.0 cm
* 18 to 50 years of age at the time of screening
* Heavy menstrual bleeding >80 mL documented by MP during the bleeding episode following the screening visit
* Normal or clinically insignificant cervical smear not requiring further follow-up
* An endometrial biopsy performed at the screening visit 1 (Visit 1), without significant histological disorder such as endometrial hyperplasia or other significant endometrial pathology
* Use of a non-hormonal barrier method of contraception starting at the bleeding episode following the screening visit 1 (Visit 1) until the end of the study
* Good general health (except for findings related to uterine fibroids)

Exclusion Criteria:

* Pregnancy or lactation
* Uterine fibroid with largest diameter >10.0 cm
* Hypersensitivity to any ingredient of the study drug
* Laboratory values outside inclusion range before randomization and considered as clinically relevant
* Hemoglobin values <6 g/dL or any condition requiring immediate blood transfusion (subjects with hemoglobin values <10.9 g/dL will receive iron supplementation)
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 309 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (92):
- United States (32):
  - Mesa, Arizona
  - Tucson, Arizona
  - San Diego, California
  - Denver, Colorado
  - Southington, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Plantation, Florida
  - South Miami, Florida
  - Sandy Springs, Georgia
  - Naperville, Illinois
  - Newburgh, Indiana
  - Marrero, Louisiana
  - Lincoln, Nebraska
  - Moorestown, New Jersey
  - Neptune City, New Jersey
  - New Brunswick, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Frisco, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle, Washington
- Belgium (4):
  - Bruxelles - Brussel
  - Charleroi
  - Leuven
  - Liège
- Bulgaria (3):
  - Pleven
  - Sofia
  - Stara Zagora
- Canada (5):
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Pointe-Claire, Quebec
  - Québec
- Czechia (5):
  - České Budějovice
  - Hradec Králové
  - Olomouc
  - Písek
  - Prague
- Finland (5):
  - Espoo
  - Helsinki
  - Joensuu
  - Kuopio
  - Oulu
- Germany (9):
  - Karlsruhe, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Geseke, North Rhine-Westphalia
  - Dresden, Saxony
  - Bernburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
  - Berlin
  - Ilsede
- Hungary (4):
  - Debrecen
  - Kecskemét
  - Szeged
  - Szentes
- Japan (12):
  - Matsudo, Chiba
  - Iizuka, Fukuoka
  - Kōriyama, Fukushima
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Ōmura, Nagasaki
  - Numazu, Shizuoka
  - Kita-ku, Tokyo
  - Nakano-ku, Tokyo
  - Tacchikawa, Tokyo
  - Kumamoto
  - Nagano
- Norway (4):
  - Nesttun
  - Oslo
  - Sellebakk
  - Trondheim
- Spain (4):
  - Aravaca, Madrid
  - Barcelona
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Örebro
  - Stockholm
  - Uppsala
- Bern, Switzerland

REFERENCES:
- [Derived] Ren X, Xia J. An algorithm for computing profile likelihood based pointwise confidence intervals for nonlinear dose-response models. PLoS One. 2019 Jan 25;14(1):e0210953. doi: 10.1371/journal.pone.0210953. eCollection 2019. PMID 30682081
- [Derived] Bradley LD, Singh SS, Simon J, Gemzell-Danielsson K, Petersdorf K, Groettrup-Wolfers E, Ren X, Zvolanek M, Seitz C. Vilaprisan in women with uterine fibroids: the randomized phase 2b ASTEROID 1 study. Fertil Steril. 2019 Feb;111(2):240-248. doi: 10.1016/j.fertnstert.2018.10.012. Epub 2018 Dec 7. PMID 30527839
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 12 countries worldwide between 15 May 2014 (first subject first visit) and 04 May 2016 (last subject last visit).
Pre-assignment Details: 748 subjects were screened; 439 subjects were not randomized, the majority was screen failures. Therefore, 309 subjects were randomized.
Groups:
- VPR 4 mg: Subjects received 4 milligram (mg) VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
- VPR 2 mg: Subjects received 2 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
- VPR 1 mg: Subjects received 1 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
- VPR 0.5 mg: Subjects received 0.5 mg VPR tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
Period: Overall Study
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Started | 62 | 61 | 63 | 62 | 61
Treated | 60 | 61 | 61 | 60 | 58
Completed Treatment | 57 | 60 | 61 | 56 | 52
Completed Follow-up | 54 | 47 | 56 | 42 | 44
Completed | 54 | 47 | 56 | 41 | 43
Not Completed | 8 | 14 | 7 | 21 | 18
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 4 | 3 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 3
Not completed — Pregnancy | 0 | 1 | 0 | 1 | 0
Not completed — Wish for pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 1 | 5 | 6
Not completed — Lost to Follow-up | 1 | 3 | 0 | 9 | 0
Not completed — Not treated | 2 | 0 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is reported for the Full Analysis Set/Safety Analysis Set (including all subjects who took at least 1 dose of study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (4.2) | 43 (4.6) | 41.9 (4.5) | 41.7 (4.9) | 42.8 (5.1) | 42.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 61 | 60 | 58 | 300
  Male | 0 | 0 | 0 | 0 | 0 | 0
Baseline menstrual blood loss by MP [Mean (Standard Deviation); unit: millilitre(s)] | 172.3 (111.86) | 176.9 (128.71) | 178.2 (116.64) | 173.6 (94.62) | 164.6 (78.71) | 173.2 (107.21)
Volume of largest fibroid by US [Mean (Standard Deviation); unit: millilitre(s)] | 78.92 (95.644) | 77.66 (91.605) | 74.55 (88.397) | 81.69 (85.62) | 99.03 (117.379) | 82.22 (95.94)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Amenorrhea, Defined as no Scheduled or Unscheduled Bleeding/Spotting After the End of the Initial Bleeding Episode Until End of Treatment
Description: Amenorrhea was defined as no scheduled or unscheduled bleeding/spotting after the end of the initial bleeding episode until end of treatment. Dose-response curve was estimated based on the primary endpoint. The 4 parameters characterizing the dose-response curve were reported in other pre-specified endpoints below.
Time Frame: After end of the initial bleeding episode until the end of treatment, up to 12 weeks
Measure: Number; unit: Percentage of subjects
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58
Percentage of subjects | 60 | 54.1 | 55.7 | 30 | 1.7
Statistical Analysis 1: Comparison: VPR 4 mg vs Placebo; The placebo-adjusted amenorrhea rate was summarized by dose with unconditional 2-sided 95% confidence intervals for each active treatment group. This unconditional confidence interval was calculated by inverting 2 separate one-sided tests of half the nominal significance level each; Test type: Superiority or Other; Percentage difference = 58.28, 95% CI 2-sided [44.55 to 70.94]
Statistical Analysis 2: Comparison: VPR 2 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage difference = 52.37, 95% CI 2-sided [38.8 to 65.42]
Statistical Analysis 3: Comparison: VPR 1 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage difference = 54.01, 95% CI 2-sided [40.41 to 66.95]
Statistical Analysis 4: Comparison: VPR 0.5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage difference = 28.28, 95% CI 2-sided [15.92 to 41.5]

2. Secondary Outcome: Change in Volume of Menstrual Blood Loss Per 28 Days From Baseline During Treatment by Reference Period (Assessed by Alkaline Hematin Method)
Description: In the below table, "N" signifies subjects who were evaluable for the specific parameter at that timepoint for each arm, respectively.
Time Frame: From baseline to end of follow-up
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58
mL
  1st period (N=46, 46, 47, 45, 45) | -79.83 (234.22) [lower limit 234.22] | -30.18 (106.82) [lower limit 106.82] | -55.42 (109.29) [lower limit 109.29] | -44.14 (110.61) [lower limit 110.61] | 17.22 (124.14) [lower limit 124.14]
  2ndperiod (N=44, 45, 47, 44, 44) | -203.43 (215.23) [lower limit 215.23] | -166.71 (149.57) [lower limit 149.57] | -181.76 (111.98) [lower limit 111.98] | -146.32 (136.97) [lower limit 136.97] | -28.42 (113.93) [lower limit 113.93]
  3rd period (N=43, 45, 47, 43, 40) | -205.08 (214.8) [lower limit 214.8] | -173.38 (153.37) [lower limit 153.37] | -185.77 (106.91) [lower limit 106.91] | -147.55 (138.4) [lower limit 138.4] | -36.69 (117.98) [lower limit 117.98]

3. Secondary Outcome: Time to Onset of Controlled Bleeding
Description: Onset of controlled bleeding was defined by the first day, for which the MBL (assessed by MP, Version 2014) for all subsequent 28-day periods up to the end of the treatment period was less than 80 mL. Kaplan-Meier estimated time to onset of controlled bleeding (days) was reported.
Time Frame: During treatment period
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 59 | 53 | 26
Days | 2 [1 to 3] | 2 [1 to 3] | 3 [1 to 3] | 2 [1 to 4] | NA [32 to NA] — insufficient number of participants with events

4. Secondary Outcome: Change in Volume of Largest Fibroid Compared to Baseline Measured by MRI
Description: Pelvic Magnetic resonance imagings (MRI), without contrast agents, were performed for volume measurements of the uterus and fibroids preferably using 1.5 Tesla scanners or higher. Images were sent to the imaging core laboratory for evaluation. Volume measurements of the uterus and fibroids were performed centrally by independent radiologist(s).
Time Frame: From baseline to end of follow-up period
Measure: Median (Full Range); unit: mL
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58
mL
  End of treatment (N=47, 52, 58, 47, 48) | -41.4 [-98 to 10] | -27.2 [-81 to 47] | -18.9 [-85 to 11314] | -14.9 [-68 to 74] | 4.9 [-67 to 271]
  Follow-up (N=45, 48, 55, 40, 41) | -26.9 [-94 to 18] | -15 [-82 to 52] | -9.7 [-79 to 437] | -9.3 [-96 to 91] | 5.1 [-59 to 364]

5. Other Pre Specified Outcome: Exposure-response Analysis of Vilaprisan - Percentage of Subjects Achieving Maximum Effect (Emax) of Induced Amenorrhea
Description: Maximum effect of vilaprisan on induced amenorrhea during treatment period. Induced amenorrhea was defined as number of subjects with amenorrhea (that is, all days with bleeding intensity 1 = none) , i.e. no bleeding or spotting allowed after initial bleeding episode until end of treatment. The nature of this exposure response analysis was the development of a model valid for the exposure response relationship over the entire range of available exposures (i.e. across all dose groups). Therefore, observations (exposure - induced amenorrhea) of all subjects need to be combined.
Time Frame: From start of the study treatment to Day 84 (treatment period)
Population: The exposure response analysis includes all verum treated subjects with valid PK concentration data and valid PD data and all placebo treated subjects with valid PD data (placebo: 50, 0.5 mg 50, 1.0 mg 56, 2.0 mg: 56, 4.0 mg: 55, in total 267).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Full Analysis Set: FAS (N=300) included all subjects who took at least 1 dose of study drug. Only subjects with valid data for this assessment were included
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 267
Percentage of subjects | 59 [49 to 68]

6. Other Pre Specified Outcome: Steady-state Exposure Achieving Half-maximal Effect (EAUC50) of Induced Amenorrhea During Treatment Period of Vilaprisan
Description: Area-under-the-curve (AUC) of vilaprisan between 0 and 24 hours post-dose at steady-state achieving 50% of maximum effect of vilaprisan on induced amenorrhea during treatment period. Induced amenorrhea was defined as number of subjects with induced-amenorrhea (that is, all days with bleeding intensity 1 = none) , i.e. no bleeding or spotting allowed after initial bleeding episode until end of treatment. The nature of this exposure response analysis was the development of a model valid for the exposure response relationship over the entire range of available exposures (i.e. across all dose groups). Therefore, observations (exposure - induced amenorrhea) of all subjects need to be combined.
Time Frame: From start of the study treatment to Day 84 (treatment period)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: mcg*h/L
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 267
mcg*h/L | 36.93 [27.69 to 48.69]

7. Other Pre Specified Outcome: Exposure-response Analysis of Vilaprisan - Predicted Percentage of Subjects Below 90% of the Maximum Probability of Induced Amenorrhea
Description: The final exposure-response model was used to simulate the percentage of subjects below 90% of the maximum probability of induced amenorrhea (that is, all days with bleeding intensity 1 = none) for the selected doses 1, 2 and 3 mg (see table below).
Time Frame: From start of the study treatment to Day 84 (treatment period)
Measure: Number; unit: Percentage of subjects
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 267
Percentage of subjects
  1 mg | 36
  2 mg | 2
  3 mg | 1

8. Other Pre Specified Outcome: Assessment of MP to Identify Subjects With Heavy Menstrual Bleeding (HMB)
Description: The ability of the MP to identify subjects with HMB (defined as > 80 mL of blood loss during bleeding episode) per 28 days against the the current gold standard (i.e. AH method) was assessed. Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of MP method for detecting heavy menstrual bleeding were calculated against AH method. Sensitivity = true positive/(true positive + false negative)*100; Specificity = true negative/(true negative + false positive)*100; PPV = true positive/(true positive + false positive)*100; NPV = true negative/(true negative + false negative)*100. MP version 2014 was originally defined based on studies in healthy subjects. And MP version 2016 was developed for study population of women with heavy bleeding.
Time Frame: At baseline
Population: An analysis set for the assessment of the interchangeability of the MP and the AH method to judge MBL included all screened subjects (except subjects in Japan) with any sanitary product data for which there is any matching pair of MP score and AH value available. A total of 399 subjects were included in this analysis set.
Measure: Number; unit: Percentage
Groups:
- Method Interchange Analysis Set: Method interchange analysis set (N=399) for the assessment of the interchangeability of the menstrual pictogram (MP) and the alkaline hematin (AH) method to judge menstrual blood loss (MBL) included subjects with sanitary product data for which there was a matching pair of MP score and AH value available.
Arm/Group | Method Interchange Analysis Set
Number analyzed (Participants) | 399
Percentage
  Version 2014: Sensitivity | 83.3
  Version 2014: Specificity | 77.3
  Version 2014: PPV | 82.1
  Version 2014: NPV | 78.7
  Version 2016: Sensitivity | 89.7
  Version 2016: Specificity | 54.5
  Version 2016: PPV | 70.6
  Version 2016: NPV | 81.4

9. Other Pre Specified Outcome: Percentage of Subjects With Amenorrhea (Defined as MBL < 2 mL) During the Last 28 Days of Treatment
Time Frame: Last 28 Days of Treatment
Measure: Number; unit: Percentage of subjects
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58
Percentage of subjects | 83.33 | 88.52 | 85.25 | 65 | 8.62

10. Other Pre Specified Outcome: Percentage of Subjects With HMB Response During the Last 28 Days of Treatment
Time Frame: Last 28 Days of Treatment
Measure: Number; unit: Percentage of subjects
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Number analyzed (Participants) | 60 | 61 | 61 | 60 | 58
Percentage of subjects | 93.33 | 96.72 | 93.44 | 81.67 | 29.31

11. Other Pre Specified Outcome: Estimated Dose-response Curve Based on Amenorrhea - E0 and Emax
Description: The primary objective was to estimate the dose-response curve based on the primary endpoint: subjects with amenorrhea. The number of subjects with amenorrhea was assumed to be binomial distributed. A 4 parameters logistic model was used to fit the observed data for characterizing the dose-response curve: E0, Emax, ED50 and δ. The model is defined as p(d)=E0 + Emax/{1+ e^[{ED50-d)/δ]}. E0 is the amenorrhea rate for placebo; Emax is the maximum effect attributable to the drug (compared with the basal effect with dose at d=0 [placebo group], the maximum increase of drug effect).
Time Frame: After end of the initial bleeding episode until the end of treatment
Measure: Number; unit: Percentage
Groups:
- Full Analysis Set: FAS (N=300) included all subjects who took at least 1 dose of study drug.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 300
Percentage
  E0 | 0.82
  Emax | 57

12. Other Pre Specified Outcome: Estimated Dose-response Curve Based on Amenorrhea - ED50
Description: The primary objective was to estimate the dose-response curve based on the primary endpoint: subjects with amenorrhea. The number of subjects with amenorrhea was assumed to be binomial distributed. A 4 parameters logistic model was used to fit the observed data for characterizing the dose-response curve: E0, Emax, ED50 and δ. The model is defined as p(d)=E0 + Emax/{1+ e^[{ED50-d)/δ]}. ED50 is the dose at which 50% of Emax were achieved.
Time Frame: After end of the initial bleeding episode until the end of treatment
Measure: Number; unit: mg
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 300
mg | 0.5

13. Other Pre Specified Outcome: Estimated Dose-response Curve Based on Amenorrhea - δ
Description: The primary objective was to estimate the dose-response curve based on the primary endpoint: subjects with amenorrhea. The number of subjects with amenorrhea was assumed to be binomial distributed. A 4 parameters logistic model was used to fit the observed data for characterizing the dose-response curve: E0, Emax, ED50 and δ. The model is defined as p(d)=E0 + Emax/{1+ e^[{ED50-d)/δ]}. δ is hill slope parameter which measures sensitivity of the response to the dose range of the drug, determining the steepness of the dose-response curve.
Time Frame: After end of the initial bleeding episode until the end of treatment
Measure: Number; unit: Slope
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 300
Slope | 0.145

ADVERSE EVENTS:
Time Frame: From start of study treatment until the end of the 6-month follow-up period
Groups:
- Placebo: Subjects matching placebo tablet once daily orally for 12 weeks (84 days) from the first week of the menstrual cycle following randomization.
Arm/Group | VPR 4 mg | VPR 2 mg | VPR 1 mg | VPR 0.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/60 | 4/61 | 3/61 | 2/60 | 2/58
Other Adverse Events (participants affected / at risk) | 31/60 | 30/61 | 31/61 | 32/60 | 32/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPR 4 mg (N=60) | VPR 2 mg (N=61) | VPR 1 mg (N=61) | VPR 0.5 mg (N=60) | Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPR 4 mg (N=60) | VPR 2 mg (N=61) | VPR 1 mg (N=61) | VPR 0.5 mg (N=60) | Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (4) | 2 (2) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (9) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (5) | 1 (1) | 2 (2) | 4 (4) | 7 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Weight increased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (8) | 5 (6) | 7 (13) | 5 (9) | 7 (11)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (5) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (3) | 4 (6) | 6 (6) | 3 (4) | 4 (6)
Metrorrhagia (Reproductive system and breast disorders) | 5 (7) | 7 (17) | 7 (10) | 4 (5) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 4 (5) | 5 (5) | 4 (6) | 15 (16) | 5 (7)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 8 (8) | 5 (5) | 5 (6) | 6 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less